CLINICAL TRIAL: NCT01212978
Title: Overcoming Inactivity in Older Adults: Impact on Vascular Homeostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Michael E. Widlansky, Assistant Professor of Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MCW-MEW2; 10GRNT3880044 (Other Grant/Funding Number: The American Heart Association)
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Aging; Cardiology; Nitric Oxide
Keywords: Aging; Endothelium,Vascular; Arterial Remodeling; Ventricular Vascular Coupling; Nitric Oxide; Walking; Software

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Delayed Intervention (No Intervention): These subjects will neither receive a pedometer or access to the motivational software until completion of the study.
- Pedometer only (Active Comparator): Participants in the this arm will receive a pedometer with instructions to reach a goal of 10,000 steps/day but will not receive access to the motivational software.
  Interventions: Behavioral: Pedometer to Increase Physical Activity
- Pedometer + Motivational Software (Experimental): In this arm, subjects will receive access to both a pedometer and motivational software
  Interventions: Behavioral: Pedometer to Increase Physical Activity

INTERVENTIONS:
Behavioral: Pedometer to Increase Physical Activity — The pedometer will be given to arms 2 and 3 (pedometer only and pedometer+software intervention) to help them guide their increase in physical activity.
  Other Names: Omron Pocket Pedometer
  Arms: Pedometer + Motivational Software; Pedometer only

SUMMARY:
The American Heart Association (AHA) and American College of Sports Medicine (ASCM) recommend older adults (50≤ age ≤ 80) perform at least 30 minutes of moderate-intensity aerobic exercise on most days ( ≥5 days) of the week. This suggestion arises, in part, from data supporting that regular physical activity reduces the risk of adverse cardiovascular events A portion of these benefits may be from reductions in the incidence and severity of cardiovascular risk factors, including diabetes mellitus, obesity, and hypertension.

While this recommendation for physical activity has been in existence for almost 15 years, the rates of obesity in the United States continue to rise and prevalence of sedentarism remains at best unchanged. Researchers have been engaged in investigating novel interventions to designed increase physical activity to reach the recommended activity targets. One promising intervention involves use of inexpensive, easy to use pedometers that allow individuals to objectively track the number of steps taken during a set period of time. Recent data suggest that an average of 10,000 steps/day as measured by a pedometer accurately estimates the activity levels recommended by the AHA, ASCM, and US government public health guidelines.

While the benefits of habitual exercise are well-documented, there are no data that demonstrate current recommendations for moderate physical activity in older adults by the ASCM, AHA, and US public health guidelines reduce the risk of adverse cardiovascular events. Interestingly, prior work indicates that pedometer-centered interventions can increase physical activity, suggesting that this type of intervention could potentially lead to cardiovascular benefits. Using validated surrogate markers of cardiovascular risk including brachial artery endothelial function, tonometric measurements of vascular stiffness, and measurements derived from transthoracic echocardiography, we will determine whether increasing the physical activity of sedentary adults to an average of 10,000 steps or more/day translates into improvements in cardiovascular health. This will be determined in the context of a randomized control trial employing a control group, a study group that uses a pedometer alone, and an intervention that couples a pedometer with internet-based motivational messaging software demonstrated in our preliminary data to encourage older adults to reach and exceed the 10,000 steps/day goal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 and ≤90 years of age
* Able to Ambulate without an Assist Device

Exclusion Criteria:

* History of Uncontrolled Diabetes Mellitus (Type 1 or 2) HgA1C >9.0%
* Uncontrolled hypertension with a blood pressure greater than 160/100 mmHg at the screening visit.
* Known history of chronic renal insufficiency, liver dysfunction, or cancer besides non-melanoma skin carcinomas or localized prostate cancer requiring systemic treatment within five years of enrollment.
* Known history of cognitive impairment or inability to follow study procedures
* History of limb amputation other than toes
* History or Reynaud's Disease
* Unable to button a shirt or blouse
* Pregnancy

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2013-07-01 (Actual)

PRIMARY OUTCOMES:
Flow induced Dilation of the Brachial Artery (FMD%) | 12 weeks

SECONDARY OUTCOMES:
Left Ventricular Systolic Performance | 12 weeks
  Ventricular systolic stiffness and arterial elastance
Left Ventricular Diastolic Function | 12 weeks
  Use of multiple echocardiographic parameters to measure

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Widlansky, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Swartz AM, Cho CC, Welch WA, Widlansky ME, Maeda H, Strath SJ. Pattern Analysis of Sedentary Behavior Change after a Walking Intervention. Am J Health Behav. 2018 May 1;42(3):90-101. doi: 10.5993/AJHB.42.3.9. PMID 29663984
- [Derived] Suboc TB, Strath SJ, Dharmashankar K, Coulliard A, Miller N, Wang J, Tanner MJ, Widlansky ME. Relative importance of step count, intensity, and duration on physical activity's impact on vascular structure and function in previously sedentary older adults. J Am Heart Assoc. 2014 Feb 26;3(1):e000702. doi: 10.1161/JAHA.113.000702. PMID 24572255